CLINICAL TRIAL: NCT00680290
Title: The Effect of Low Intensity Exercise on Quality of Life and Hemodynamics in Patients With Permanent Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTSW IRB 072004-047
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation
Keywords: exercise, quality of life, cpx
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity; Coproporphyria, Hereditary | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Exercise group
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — Exercise x 8 weeks

SUMMARY:
The purpose of this study is to 1) assess the effect of routine exercise on the quality of life of patients with permanent atrial fibrillation, and 2) assess the effect of exercise on cardio-hemodynamics in patients with atrial fibrillation.

DETAILED DESCRIPTION:
1. Twelve patients will be enrolled. Each subject will first serve as their own control and then serve in the treatment group. Subjects will be required to sign informed consent prior to any study procedure.
2. The exercise program will be structured as follows:

   At the time of enrollment, patients will undergo an exercise treadmill test to measure cardiac hemodynamics, including VO2max (measured non-invasively using gas exchange) and maximal heart rate. Average heart rate over 24 hours will also be measured by a 24-hour Holter monitor before and after the exercise program. The maximal exercise testing will be performed on a treadmill using an incremental protocol based on the estimated fitness level established during a warm up.

   For the first 8-weeks of their participation, patients will act as their own control and not exercise. When the 8 week period is complete, they will return for another exercise treadmill test and 24-hour Holter monitor.

   For the second 8-weeks of their participation, patients will participate in exercise training. The initial 2 weeks of exercise will be supervised at the St. Paul University Hospital exercise facility for twenty minutes a day, four times a week. Exercise will be done by walking or use of aerobic exercise equipment, which include a treadmill, elliptical machine, cycle ergometer or rowing machine according to patient preference and availability of exercise facilities at home.

   During this period the patients will commence training at an intermediate effort based on perceived exertion (Borg Scale 11-13). The intensity will be gradually increased to a level corresponding to 70-75% VO2max or 15 on the Borg Scale, whichever represents the least effort.

   For the remaining six weeks, the patients will continue the exercise program at the perceived intensity learned during the first two weeks of training. During these six weeks, the patients will be asked to exercise for 30 minutes, five times per week.

   Participants can exercise at home if they wish, but they will be required to undergo supervised exercise at least once per week during this six week period and will be required to keep an exercise log for monitoring their unsupervised efforts.

   At the end of this 8-week program of exercise training, patients will return for a third exercise treadmill test and 24-hour Holter monitor.
3. The Quality of Life survey will be assessed with two forms, the Short Form 36 (SF 36) and the Arrhythmia Related Symptom Severity Check List (SSCL). Patients will be asked to fill out both the SF 36 QOL and SSCL QOL survey and submit to a Physical Activity Recall (PAR) interview each time they have the exercise treadmill test and 24-hour Holter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with permanent atrial fibrillation for at least three months duration, on stable medical therapy and in whom no additional interventions are planned to treat AF either due to clinical reasons or patient preferences
2. Have the ability to understand and sign consent to participate and be willing and able to comply with prescribed exercise and schedule of evaluations
3. Sedentary lifestyle as determined by Physical Activity Recall (PAR)
4. Be greater than 18 years of age

Exclusion Criteria:

1. Inability to exercise
2. Functional Class IV CHF symptoms
3. Active symptoms of angina, coronary artery disease
4. Patient with recent history of myocardial infarction
5. Patient with moderate or severely depressed left ventricular function (LVEF < 40 %)
6. Patient with any significant co-morbidities that may limit ability to exercise
7. Patients already engaged a structured exercise program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
to 1) assess the effect of routine exercise on the quality of life of patients with permanent atrial fibrillation, and 2) assess the effect of exercise on cardio-hemodynamics in patients with atrial fibrillation. | 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Joglar, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States